CLINICAL TRIAL: NCT01123993
Title: The Effect of Thai Traditional Music on Cognitive Function, Psychological Health and Quality of Sleep Among Thai Older Individuals With Dementia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Dr.Pasiri Sithinamsuwan, Neurologist staff, Division of Neurology, Department of medicine, Phramongkutklao Hosptial and College of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R006h/53
Record Dates: First submitted 2010-05-02; First posted 2010-05-14 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2011-01

CONDITIONS: Cognitive Function; Sleep
Keywords: Thai traditional music; dementia; Cognitive function; behavioural problem; sleep quality; psychological health; quality of sleep
MeSH Terms: conditions — Dementia; Mental Disorders; Sleep Initiation and Maintenance Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle counselling (No Intervention)
  Interventions: Device: Music CD

INTERVENTIONS:
Device: Music CD — During 4-week interventional period of each group, a researcher gives a CD to care giver and advises him/her to open the music for patient for at least 60 minutes daily, after dinner to bedtime. Meanwhile, the care giver notes the exact duration that patient actually listens to it in the calendar provided and returns the CD and document to the researcher at the end of interventional period.

SUMMARY:
To determine the effect of Thai traditional music on cognitive function, psychological health and quality of sleep among Thai older individuals with dementia.

DETAILED DESCRIPTION:
Dementia, regardless of its cause, has been recognized to be one of the most important and common problems among the elderly worldwide. The prevalence of dementia has been increasing gradually throughout the world. It is associated with medical and psychological consequences, especially in the advanced stage of the condition. Medications for dementia, specifically, acetylcholine esterase inhibitors, have proven efficacy but variable individual response. They are very expensive and stress families and insurance payers. Dementia and its neuropsychiatric co-morbidities effects not only individual patients, but also family members and care givers as it stresses interpersonal relationships, increases the need for personal care, nursing home placement, and the use of neuropsychiatric medications. Any new approach to improve cognitive function, behavior, mood and sleep quality among demented individuals therefore could have far reaching benefits for patients, care givers, financially responsive parties, and the country as a whole.

There are several studies focusing on the non-pharmacologic approaches to care of the demented. The objectives were to reduce reliance on prescribed medications with these adjunctive therapies. One of the interesting non-drug trials was about music therapy. It was found that music could improve behavioral and social functions among individual demented patients. However, the methodology of each music study varied considerably. To our knowledge, there has been no music study in dementia performed in Thailand using our unique Thai traditional music. We therefore aim to study this non-pharmacologic approach in Thai demented individuals using Thai traditional music. We hypothesized that regular listening to Thai traditional music will improve cognitive function, activities of daily living, mood, behavior and sleep quality in Thai demented patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years
* Diagnosed with Alzheimer's disease, vascular dementia or mixed dementia by ICD-10
* No change in neuropsychiatric drugs for at least 4-week before and 8-week during the study
* CD player available at home
* Patient and care giver consent to study

Exclusion Criteria:

* Severe depression requiring aggressive treatment or hospitalization
* Dementia with Lewy body, multisystem atrophy
* Treatable dementia
* Active medical problems
* Profound hearing loss

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Depression | 4-week after regularly listening to the music for 28 days
  Using Thai Geriatric Depression Scale (TGDS)
Activities of Daily Living | 4-week after music
  using AD Cooperative Study Activities of Daily Living Inventory (ADCS/ADL)
Behavior | 4-week after music
  Using Behavioral pathology in Alzheimer's Disease Rating Scale (BEHAVE AD)
Sleep quality | 4-week after music
  Using Pittsburgh Sleep Quality Index (PSQI)

SECONDARY OUTCOMES:
reduction of the care giver's stress and burden | 4-week after intervention
  Using visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Pasiri Sithinamsuwan, MD, Principal Investigator — Neurologic Clinic, Division of Neurology, Department of Medicine, Phramongkutklao Hospital, Bangkok, 10400, Thailand; Sansanee Saengwanitch, MD, Study Chair — Neurologic Clinic, Division of Neurology, Department of Medicine, Phramongkutklao Hospital, Bangkok, 10400, Thailand; Thanawong Yongarnukul, Study Chair — Phramongkutklao College of Medicine; Tanuphat Tuan-iam, Study Chair — Phramongkutklao College of Medicine; Kanokporn Wonganankit, Study Chair — Phramongkutklao College of Medicine; Chananya Potisuk, Study Chair — Phramongkutklao College of Medicine; Sittichoke Sirimontakan, Study Chair — Phramongkutklao College of Medicine; Sariya Wongsangsak, Study Chair — Phramongkutklao College of Medicine; Akarachaid Pinidbunjerdkool, MD, Study Chair — Neurologic Clinic, Division of Neurology, Department of Medicine, Phramongkutklao Hospital, Bangkok, 10400, Thailand; Mathirut Mungthin, MD, Study Director — Phramongkutklao College of Medicine
Locations (2):
- Thailand (2):
  - Neurologic Clinic, Division of Neurology, Department of Medicine, Phramongkutklao Hospital, Bangkok, Bangkok
  - Division of Neurology, Phramongkutklao Hospital, Rachatevee, Bangkok